CLINICAL TRIAL: NCT04139876
Title: Ligasure Hemorrhoidectomy Versus Open Hemorrhoidectomy. A Randomized Clinical Trial on the Long-term Effect on Hemorrhoidal Symptoms
Brief Title: Ligasure Hemorrhoidectomy Versus Open Hemorrhoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, André Heiner dos Santos Campos, MD, Holbaek Sygehus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Holbaek
Record Dates: First submitted 2019-10-04; First posted 2019-10-25 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoidectomy; Minimal Open hemorrhoidectomy; LigaSure hemorrhoidectomy
MeSH Terms: conditions — Hemorrhoids | interventions — Hemorrhoidectomy

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal open hemorrhoidectomy (Active Comparator): Patients randomized to Minimal open hemorrhoidectomy
  Interventions: Procedure: Open Haemorrhoidectomy
- LigaSure hemorrhoidectomy (Active Comparator): Patients randomized to LigaSure hemorrhoidectomy
  Interventions: Procedure: LigaSure Hemorrhoidectomy

INTERVENTIONS:
Procedure: Open Haemorrhoidectomy — Patient operated in the lithotomy position. The external components are grasped by clamps using gentle traction. Diathermy is used for dissection and hemostasis. The skin is incised midway to one-third of the distance from the top of the pedicle, thus, minimizing the skin excision. The subdermal fascia continuing into a submucosal fascia covering the internal anal sphincter is identified as are fibers passing between the hemorrhoid (H) and this fascia. The H is dissected free from the underlying internal sphincter in this plane, leaving the sphincter unharmed. The anal mucosa is incised at the transition from anal mucosa to hemorrhoidal mucosa and only anal mucosa overlying the H is excised. Only the caudal part of the H is excised. With the H held with gentle traction it is divided at the anal orifice. There will thus be a residual part of the H intra-anally with its caudal end 1-2 cm proximal to the anal orifice.
  Other Names: Milligan Morgan; Minimal open Hemorrhoidectomy; Hemorrhoidectomy
  Arms: Minimal open hemorrhoidectomy
Procedure: LigaSure Hemorrhoidectomy — Patient is operated in the lithotomy position. The main haemorrhoidal (H) masses are identified and delineated. The H are prolapsed out from the anal canal with Allis clamps or similar pick up forceps. Tension is applied to visualise the junction between the nodule and the mucosal wall (internal) or the perianal tissue (external). A small V-shaped anodermal seal is performed by applying the LigaSure (LS) forceps close to the edge of each pile. The seal is then transacted with scissors along the line of coagulum. Care should be taken to limit the amount of tissue removed to minimize the stricture risk. Repeated applications of the device are performed and the excision is continued into the anal canal, lifting the pile from the internal anal sphincter to the level of the vascular pedicle that is finally sealed by LS and divided.
  Arms: LigaSure hemorrhoidectomy

SUMMARY:
This is a single center randomized clinical trial comparing Ligasure Hemorrhoidectomy and Open Hemorrhoidectomy for the treatment of prolapsing haemorrhoids. The primary aim of the study is to evaluate symptoms related to hemorrhoids one year postoperatively, according to a hemorrhoidal disease symptom score (HDSS).

Secondary endpoints are patient satisfaction with the operation, Health related Quality of Life and effect on anal continence.

DETAILED DESCRIPTION:
Background

Hemorrhoids is one of the oldest known medical conditions. Description of hemorrhoids is found as early as 2250 Before Christ (BC) in the code of king Hammurabi in Babylon. Even though first recorded treatment is thought to be found in the "Edwin Smith Papyrus" from 1700 BC as of today the treatment of this benign state is still debated. A wide range of prevalence rates of hemorrhoids have been stated in part because of the varying definition ,but the general consensus is that hemorrhoidal disease is a common anorectal disease affecting the quality of life of millions of people worldwide. Operation for hemorrhoid is one of the most common operations for benign disease in Denmark.

Hemorrhoids arise from the normal vascular structures in the anal canal also referred to as anal cushions or sinusoids as they do not contain muscular cells like arteries or veins. These cushions are typically arranged in three main columns or piles in the anal canal forming an important part of the intricate mechanism of the anal canal preventing incontinence.

Hemorrhoids is a pathologic term describing the symptomatic abnormal downward displacement and enlargement of the anal cushions. The term hemorrhoidal disease is used when the hemorrhoids cause symptoms.

Treatment of hemorrhoidal disease consists of conservative management with lifestyle and diet changes or local treatment, minor surgery and surgical treatment depending on the severity of disease and symptoms. The staging of internal hemorrhoids in four categories by the Goligher classification is the classification that generally forms the basis of the treatment in Denmark.

Local treatment consists of corticosteroids and anaesthetic ointments. Minor surgery includes rubber band ligation and sclerotherapy. Operation is reserved for subjects with prolapse, Goligher grade II and IV. Grade II hemorrhoids may be treated by operation if still symptomatic after banding or sclerosing.

The gold standard in the operative treatment of hemorrhoidal is the Milligan-Morgan Hemorrhoidectomy also referred to as hemorrhoidal excision or Open Hemorrhoidectomy (OH). The operation can also be performed as a Closed Hemorrhoidectomy when the wound is closed with sutures (Ferguson's Hemorrhoidectomy).

The conventional excisional operation has been associated with postprocedural pain and delayed healing of wounds. In recent years there have been suggestions for and a development toward a less traumatic Open Hemorrhoidectomy. Injuries to the internal anal sphincter during dissection is thought to be one cause for pain. The less traumatic operations include dissection of the hemorrhoid preserving the fascia over the internal anal sphincter and also smaller excision of skin and mucosa - the technique used in this study is described in more detail under Methods.

Several new procedures have been proposed in the last decades. Common for all is the implementation of a new technical device, meaning increased operative costs.

LigaSure Trademark (TM) hemorrhoidectomy (LH) is a hemorrhoidectomy performed with the use of the LigaSure TM instrument in stead of the traditional diathermy. The LigaSure TM technology patented in 1998 as "Energy Delivery System for Vessel Sealing" creates vessel fusion by a combination of pressure and energy17. The LigaSure device excises the hemorrhoids and seals the wound in the same procedure delivering the energy in a controlled way between the diathermy forceps theoretically limiting thermal spray and tissue charring.

Rationale

Hemorrhoidal Disease is a benign disease and should be evaluated by it's effect on hemorrhoidal symptoms together with its effect on quality of life.

Hemorrhoidal symptoms should be the main outcome variable when evaluating surgery for hemorrhoidal disease. This information is largely lacking.

The use of a validated symptom score with long term follow-up could yield important information for the choice of treatment of haemorrhoidal disease.

ELIGIBILITY:
Inclusion Criteria:

* The patient has Grade III-IV haemorrhoids or Grade II haemorrhoids with bleeding resistant to rubber band ligation or sclerotherapy
* The patient has a Haemorrhoidal Symptom Score of 4 or more
* The patient has an American Society of Anaesthesiologists (ASA) score I-II
* The patient's age is 18-85 years at inclusion
* The patient has had a colonoscopy, sigmoidoscopy or rigid rectoscopy within 3 months before inclusion

Exclusion Criteria:

* The patient has had previous operation for haemorrhoids within the last 2 years
* The patient has had previous operation for anal incontinence
* The patient has an active anal fistula
* The patient has an active anal fissure
* The patient has anal incontinence for solid stools
* Active immunosuppressive therapy (increased risk of anorectal sepsis)
* Cirrhosis / portal hypertension
* Mb Crohn.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Hemorrhoidal symptoms assessed by the Hemorrhoidal Disease Symptom Score (HDSS). | 1 year postoperatively
  The HDSS consists of five items on patient-reported frequency of pain, itching, bleeding, soiling and prolapse. Each symptom graded on a five-point scale (0=never, 1=less than once a month, 2=less than once a week, 3=1-6 days per week, 4=every day / always), giving a total score ranging from 0-20. Zero meaning no symptoms. (See reference).

SECONDARY OUTCOMES:
Patient satisfaction assessed by a seven grade Likert Scale. | Preoperatively (baseline) and 1 year postoperatively
  At follow-up patients grade their satisfaction with the operation on a seven-point Likert scale (1= very unsatisfied, 7 = very satisfied).
Hemorrhoidal affection of the patient's daily life assessed by Short Health Scale adapted to hemorrhoidal disease (SHSHD). | Preoperatively (baseline) and 1 year postoperatively
  SHSHD consist of four questions graded on a 7-point Likert scale. The questions deal with how the patients symptoms caused by hemorrhoids affect the patients daily life.
  1. - Overall symptom load (1 = no symptoms, 7 = severe symptoms),
  2. - Interference with daily activities (1 = not at all, 7 = interfere to a very high degree)
  3. - Worries caused by HD (1 = no concerns, 7 = constant concerns)
  4. - General well-being (1 = very good, 7 = very bad) The points of each question are summed giving a total score ranging from 4 to 28. (See reference).
Anal continence (gas and solids) assessed by the Wexner incontinence scale. | Preoperatively (baseline) and 1 year postoperatively
  Wexner incontinence scale consists of five questions on fecal incontinence graded on a five-point Likert scale from 0 to 4.
  The points of each question are summed giving a total score ranging from 0 to 20. Zero meaning no incontinence and 20 complete incontinence.
Fecal continence assessed by the Revised Fecal Incontinence Scale (RFIS). | Preoperatively (baseline) and 1 year postoperatively
  RFIS consists of five questions on fecal incontinence graded on a five-point Likert scale from 0 to 4. The points of each question are summed giving a total score ranging from 0 to 20. Zero meaning no fecal incontinence and twenty total fecal incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Per Olov Gunnar Olaison, MD, pHD, Study Director — Department of Surgery, Holbaek County Hospital
Locations (1):
- Departement of Surgery, Holbaek County Hospital., Holbæk, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rorvik HD, Styr K, Ilum L, McKinstry GL, Dragesund T, Campos AH, Brandstrup B, Olaison G. Hemorrhoidal Disease Symptom Score and Short Health ScaleHD: New Tools to Evaluate Symptoms and Health-Related Quality of Life in Hemorrhoidal Disease. Dis Colon Rectum. 2019 Mar;62(3):333-342. doi: 10.1097/DCR.0000000000001234. PMID 30451751

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT04139876/Prot_SAP_000.pdf